CLINICAL TRIAL: NCT01984021
Title: Evaluation of the Immediate Effect of Acupuncture on Pain, Cervical Range of Motion and Electromyographic Activity of the Upper Trapezius Muscle in Patients With Nonspecific Neck Pain: Randomized, Single-blinded, Sham-controlled Study.
Brief Title: Evaluation of the Immediate Effect of Acupuncture on the Upper Trapezius Muscle in Patients With Nonspecific Neck Pain.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, MSc, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 483712
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Nonspecific Neck Pain
Keywords: Physical Therapy Modalities; Neck pain; Acupuncture
MeSH Terms: conditions — Neck Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- traditional acupuncture (tACP) (Experimental): In the upper trapezius muscle with the greatest area pain and lowest PPT score will be chosen for acupuncture. Sterile acupuncture needles measuring 0.25 x 13 mm (Suzhou Huanqiu Acupuncture Medical Appliance Co. Ltd.®) will be inserted in TE-5 (located on the dorsal face of the forearm between the radius and ulna 3 cm above the joint line of the wrist) and LI-11 (located at the outermost point of the skinfold of elbow flexion in the direction of the lateral epicondyle of the elbow).
  Interventions: Device: Acupuncture
- sham acupuncture (sACP) (Placebo Comparator): The needles will be inserted 1 cm to the side of TE-5 (located on the dorsal face of the forearm between the radius and ulna 3 cm above the joint line of the wrist) and 1 cm to the side of LI-11 (in the direction of the styloid process of the radius).The acupuncture needles are positioned at different acupoints.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acupuncture
  Arms: traditional acupuncture (tACP)
Device: Sham acupuncture
  Arms: sham acupuncture (sACP)

SUMMARY:
The aim of the proposed study is to evaluate the immediate effect of acupuncture on pain, cervical range of motion and electromyographic activity of the upper trapezius muscle in patients with nonspecific neck pain.Twelve patients with nonspecific neck pain and 12 healthy subjects will be enrolled in a randomized, single-blind, crossover study. Each patient will receive two forms of treatment in random order: a single session of traditional acupuncture and sham acupuncture. To eliminate carry-over treatment effects, a one-week wash-out period will be respected between sessions. Surface electromyography will be used to determine motor control in the upper trapezius muscle before and after treatment. The outcome measures in the group with neck pain will be a numerical pain rating scale (range: 0 [no pain] to 10 [maximum pain]), documentation of the pain area on a body chart and cervical range of motion. Linear regression analysis will be applied for each individual to investigate associations between the sEMG variables and force (excluding the sixth step). The slopes of the regression lines will be used to measure the sensitivity of the sEMG variables regarding changes in force. The Shapiro-Wilk test will be used to test the normality of the data distribution regarding RMS and MDF values in the third and sixth step of the step contraction. Paired samples (Student's t-test or Wilcoxon test) will be used to test differences between third and sixth contraction step. A mixed linear model will be used to analyze and compare the sEMG data during sustained contraction (five steps) between pre-acupuncture (EMG-1) and post-acupuncture (EMG-2) evaluations. These comparisons will demonstrate whether acupoints TE-5 and LI-11 affect the activity of the upper trapezius muscle, as hypothesized. The pain (NRS, PPT and area) and cervical ROM data collected during the four evaluations will also be compared using a mixed linear model. The Statistical Package for Social Sciences (SPSS, version 19.0 for Windows) will be employed for the statistical analysis, with the level of significance set to 5% (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years
* male and female volunteers

Exclusion Criteria:

* history of neurological disorders
* neck surgery
* chronic neck pain resulting from a traumatic incident
* chronic musculoskeletal condition
* medical diagnosis of fibromyalgia; systemic disease
* connective tissue disorder
* non-tolerance of needles; current pregnancy
* having undergone physical therapy use of analgesic, muscle relaxant.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
electromyographic activity | 1 Year
  The EMG signal will be recorded in the dominant upper trapezius muscle in patients with nonspecific neck pain, will be evaluated before and after treatment.

SECONDARY OUTCOMES:
cervical range of motion | 1 Year
  A cervical range of motion instrument will be used to determine cervical spine movements. This instrument is composed of two gravity goniometers and a compass goniometer and has demonstrated to be a reliable tool with adequate validity. The device will be placed on the top of the head and the patient will be instructed to move the head as far as possible without pain in a standard fashion: right rotation, left rotation, flexion, extension, right lateral flexion and left lateral flexion. Three trials will be conducted in randomized order for each direction of movement and mean values will be recorded for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Calamita SA, Biasotto-Gonzalez DA, De Melo NC, dos Santos DM, de Lassa R, de Mendonca FS, Oliveira CS, Amorim CF, Gonzalez TO, Fumagalli MA, de Gomes CA, Politti F. Evaluation of the immediate effect of acupuncture on pain, cervical range of motion and electromyographic activity of the upper trapezius muscle in patients with nonspecific neck pain: study protocol for a randomized controlled trial. Trials. 2015 Mar 19;16:100. doi: 10.1186/s13063-015-0623-3. PMID 25872667
- See also: Related Info — http://www.uninove.br